CLINICAL TRIAL: NCT01880762
Title: Research Evaluation of PET/MR and PET/CT Imaging for Bone Marrow Lesions
Brief Title: Evaluation of PET/MR and PET/CT Imaging for Bone Marrow Lesions
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: S12-02920
Record Dates: First submitted 2013-03-11; First posted 2013-06-19 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Multiple Myeloma; Disease of the Marrow; Osteoporosis
Keywords: PET MR development and validation
MeSH Terms: conditions — Multiple Myeloma; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Developing an MRI protocol at 1.5 T allowing quantification of the hematopoietic, fatty and trabecular moieties of marrow. An ideal protocol would differentiate red marrow from neoplastic cellular infiltration, and detect loss of trabecular bone. This study assesses the feasibility of a multiple gradient echo sequence for differentiation of water and fat constituents of marrow, combined with T2* mapping to interrogate the trabecular component The investigators hypothesize that these techniques will allow better identification of lesion type than routine MR sequences, and can be used to quantitatively characterize myelomatous marrow replacement, with iliac crest biopsy (which is routinely performed in the diagnosis of myeloma) as gold standard.

Fluoro-deoxyglucose (FDG)/PET CT imaging can detect FDG uptake in active myeloma and is obtained routinely for certain cohorts of patients with myeloma. PET/CT is commonly used in both initial whole body assessment and in monitoring remission. PET has been found to be about 59% sensitive and 75% specific for detection of myeloma .

Myelomatous lesions are detected on MRI by the replacement of marrow fat. Routine MRI however is limited by scope/field of view, usually evaluating marrow in a single anatomic region (such as an extremity, the pelvis or spine). To assess the diffuse marrow involvement in MM, whole body MRI imaging potentiates near global assessment of the marrow, which aids in evaluating tumor burden, and may be useful in staging.

DETAILED DESCRIPTION:
Imaging of the pelvis and bilateral femora at 1.5 Tesla in a 30 minute research time "slots" at NYU-FPO MRI, Tisch Hospital, NYU Medical Center, Department of Radiology, HCC basement. This protocol utilizes routine, Dixon sequences and multi-echo MR "spectroscopic" sequences, allowing quantization of the fat water and trabecular moieties of marrow. The opposed phase portion of a Dixon sequence can aid differentiation between dense red marrow and a metastatic deposits by assaying for intravoxel fat. Diffusion sequences may also potentially improve specificity by assessing mobility of water in hypercellular and hypocellular portions of marrow, and will be added to the protocol if scan time permits.

The new sequences conform to FDA safety regulations regarding static magnetic field, time varying magnetic fields, specific absorption rate, and acoustic noise levels. However, since they have not been fully validated for diagnostic accuracy, the resulting images will be analyzed for research purposes only and will not be used in the patient's diagnostic assessment.

ELIGIBILITY:
Inclusion Criteria

* subjects who are schedule for PET CT
* subjects that are diagnosed with Multiple Myeloma.
* Healthy subjects will be enrolled to optimize imaging techniques
* subjects 30 - 80 years of age

Exclusion Criteria:

Exclusion criteria include all patients who are contraindicated for MR imaging in general.

Contraindications include:

* electrical implants such as cardiac pacemakers or perfusion pumps
* ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants
* ferromagnetic objects such as jewelry or metal clips in clothing
* pregnant subjects
* pre-existing medical conditions including a likelihood of developing seizures or claustrophobic reactions, and any greater than normal potential for cardiac arrest.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Multiple Myeloma and that are referred for PET CT imaging.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2013-01; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To Improve specificity of Multiple Myeloma using PET MR | 2 years
  WHOLE BODY MRI/PET imaging for global assessment of the marrow in patients with MM. This will determine the feasibility of a multiple gradient echo sequence for differentiation of water and fat constituents of marrow, combined with T2* mapping to interrogate the trabecular component which would allow for increased identification of lesion type than routine MR Sequences, and can be used to quantitatively characterize myelomatous marrow replacement with the current biopsy as gold standard.

SECONDARY OUTCOMES:
Newly developed MRI imaging sequences | 2 years
  New imaging sequences developed will further improve specificity and assessment of marrow diseases in multiple myeloma patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra L Moore, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Center for Biomedical Imaging, New York, New York, United States